CLINICAL TRIAL: NCT06418542
Title: Assessment of the Frequency of Fundus Fluorescein Angiography Relationship With Contrast Nephropathy and Associated Factors
Brief Title: Contrast Nephropathy Associated FFA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, NUR SENA ÇOBAN, Assistant Doctor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E-48865165
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Contrast-induced Nephropathy; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- END (Other): patients who have chronic renal disease
  Interventions: Device: use of florescein
- END free (Other): patients who don't have chronic renal disease
  Interventions: Device: use of florescein

INTERVENTIONS:
Device: use of florescein — Fluorescein, an organic contrast agent, is used in FFA to detect retinal pathologies.

SUMMARY:
After the use of iodinated contrast agents, there is a risk of developing contrast nephropathy. Limited data in the literature are available on the incidence of contrast nephropathy after fluorescein angiography (FFA), which is an iodine-free organic contrast. Additionally, factors associated with contrast nephropathy after FFA are not clearly understood. Our study aims to evaluate these points.

DETAILED DESCRIPTION:
It is known that patients are at risk of developing contrast nephropathy after FFA with iodinated contrast media. However, although it is known that contrast nephropathy may develop after FFA with fluorescein, a non-iodinated organic contrast agent, there is very limited data in the literature.

In this study, we aimed to determine the incidence of contrast nephropathy after FFA for retinopathy evaluation and to evaluate the associated factors (age, gender, diabetes mellitus, hypertension, chronic kidney disease, baseline renal function, medications, etc.). Our study was planned prospectively. Patients over the age of 18 years who applied to Prof. Dr. Cemil Taşcıoğlu City Hospital Eye Clinic as outpatients and who did not meet the exclusion criteria and agreed to participate in the study will be included in our study. Age, gender, demographic, clinical and laboratory data of these patients will be recorded from the patient file and hospital data processing system. The definition of contrast nephropathy is defined as an increase in serum creatinine (SCr) ≥0.5 mg/dL or more than 25% of the baseline value in the study titled "Contrast-induced Kidney Injury:Focus on Modifiable Risk Factorsand Prophylactic Strategies", "Risk of nephropathy after intravenous administration of contrast material: a critical literature analysis. In this study, an increase of 0.3 mg/dL in serum creatinine within 48 hours after contrast was accepted. The definition of contrast nephropathy will be evaluated separately as both an increase of 0.5 mg/dl or 25% increase in creatinine value compared to baseline and an increase of 0.3 mg/dl compared to baseline. In this way, there are studies in which the frequency of contrast nephropathy was evaluated separately according to both criteria in the same study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old. Patients with an indication for FFA. Those who agreed to participate in the study.

Exclusion Criteria:

* Patients with nephrotoxic drug exposure in the last two weeks
* Patients who underwent imaging management requiring the use of other contrast agents in the last month (such as coronary angiography, CT angiography)
* Patients with unstable hemodynamics
* Patients with obstructive uropathy
* Patients with end-stage renal failure with eGFR<15
* Patients on a routine hemodialysis program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Contrast Nephropathy associated FFA | 48-72 hours
  Urea and creatinine values will be measured 48-72 hours after FFA . The renal function of these patients one month before FFA will be compared with the renal function 48-72 hours after FFA and the development of contrast nephropathy will be determined based on KDIGO and AKIN criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided